CLINICAL TRIAL: NCT06198595
Title: Comparison of the Effectiveness of Treatments in Carbon Monoxide Intoxications: A Prospective, Observational Study
Brief Title: Comparison of the Effectiveness of Treatments in Carbon Monoxide Intoxications
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-23-5424
Record Dates: First submitted 2023-12-11; First posted 2024-01-10 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Carbon Monoxide Poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normobaric oxygen therapy group: "Patients Receiving Oxygen from Hospital Circuits at Normal Atmospheric Pressure"
- Noninvasive mechanical ventilation group: "Patients Receiving High PEEP Oxygenation Without Advanced Airway via Mechanical Ventilation"
- EzPAP Positive Airway Pressure System: "Patients Receiving Positive Airway Pressure Support for Lung Expansion Without Advanced Airway via the EzPAP Device."

SUMMARY:
Carbon monoxide (CO) poisoning is a condition that occurs as a result of inhaling carbon monoxide gas and can potentially lead to serious health issues. The treatment of CO poisoning requires urgent medical intervention. Methods used in the treatment of CO poisoning include normobaric oxygen (oxygen at normal pressure), high-flow oxygen, non-invasive continuous positive airway pressure (CPAP), and hyperbaric oxygen therapy. Studies on these methods are available in the literature.

DETAILED DESCRIPTION:
When examining the mechanisms of application for these methods:

Normobaric Oxygen Therapy: In normobaric oxygen therapy, researchers treat participants with normobaric (sea level) oxygen. This method provides high concentrations of oxygen, allowing better oxygen saturation of the blood and faster removal of carbon monoxide from the body. Participants inhale normobaric oxygen through devices such as masks or nasal cannulas.

High-Flow Oxygen Therapy: In high-flow oxygen therapy, researchers treat participants with high-flow oxygen. Typically, a nasal cannula or oxygen mask is used. The high flow rate allows more oxygen to reach the alveoli and bind to hemoglobin. This method can be effective, especially in more severe cases of carbon monoxide poisoning.

Non-Invasive CPAP Therapy: Non-invasive CPAP therapy is typically used to treat respiratory problems such as sleep apnea but can also be used in the treatment of CO poisoning. Participants receive oxygen under continuous positive airway pressure with the help of a mask.

Comparison of these methods:

Normobaric oxygen is considered the standard treatment for CO poisoning and generally effectively eliminates carbon monoxide from the body. High-flow oxygen may be more effective in providing additional oxygen in more severe cases, but it works similarly to normobaric oxygen. The choice of which treatment method to use can vary depending on the participant's clinical condition, the severity of poisoning, and other factors. The researchers main goal in designing this study is to determine which treatment, depending on the researcher's decision, most rapidly shortens the half-life of carbon monoxide in participants experiencing severe carbon monoxide poisoning.The researchers aim to identify which treatment participants tolerate better and which method minimizes complications related to CO intoxication.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65,
* Without any underlying health conditions,
* Diagnosed with carbon monoxide poisoning,
* Capable of providing consent either personally or through a legal representative.

Exclusion Criteria:

* Under the age of 18,
* Over the age of 65,
* With underlying health conditions,
* Without a diagnosis of carbon monoxide poisoning,
* Patients who do not wish to share their data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who present to the emergency department with or are brought in due to CO intoxication will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Carboxyhemoglobin | 6 hours later
  Blood carboxyhemoglobin saturation is typically expressed as a percentage. For example, the statement "blood carboxyhemoglobin saturation is 5%" indicates that 5% of hemoglobin has been converted to carboxyhemoglobin. This ratio affects the oxygen-carrying capacity of the blood and serves as an indicator of carbon monoxide poisoning. After treatment, a decrease in this ratio signifies the elimination of carbon monoxide from the body and the restoration of normal oxygen-carrying function.
lactate | 6 hours later
  Blood lactate levels are typically measured in millimoles per liter (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: SAFA DÖNMEZ, MD, Principal Investigator — ANKARA BİLKENT CİTY HOSPİTAL
Locations (1):
- Ankara Bilkent Şehir Hastanesi, Ankara, Çankaya, Turkey (Türkiye)

REFERENCES:
- [Background] Akkan S, Uyanik O. Comparing high-flow nasal oxygen therapy and normobaric oxygen therapy on the treatment of carbon monoxide poisoning. Med Klin Intensivmed Notfmed. 2024 Apr;119(3):214-219. doi: 10.1007/s00063-023-01044-5. Epub 2023 Aug 2. PMID 37530814
- [Background] Kim YM, Shin HJ, Choi DW, Kim JM, Lee SW, Jeong SH, Kim H. Comparison of high-flow nasal cannula oxygen therapy and conventional reserve-bag oxygen therapy in carbon monoxide intoxication: A pilot study. Am J Emerg Med. 2020 Aug;38(8):1621-1626. doi: 10.1016/j.ajem.2019.158451. Epub 2019 Nov 6. PMID 31706658
- [Background] Ozturan IU, Yaka E, Suner S, Ozbek AE, Alyesil C, Dogan NO, Yilmaz S, Pekdemir M. Determination of carboxyhemoglobin half-life in patients with carbon monoxide toxicity treated with high flow nasal cannula oxygen therapy. Clin Toxicol (Phila). 2019 Jul;57(7):617-623. doi: 10.1080/15563650.2018.1540046. Epub 2019 Jan 28. PMID 30689450
- [Background] Turgut K, Yavuz E. CPAP versus HFNC use in carbon monoxide poisoning. Am J Emerg Med. 2021 Aug;46:727. doi: 10.1016/j.ajem.2020.09.085. Epub 2020 Oct 2. No abstract available. PMID 33036847
- [Background] Roth D, Mayer J, Schreiber W, Herkner H, Laggner AN. Acute carbon monoxide poisoning treatment by non-invasive CPAP-ventilation, and by reservoir face mask: Two simultaneous cases. Am J Emerg Med. 2018 Sep;36(9):1718.e5-1718.e6. doi: 10.1016/j.ajem.2018.05.066. Epub 2018 May 29. PMID 29866417
- [Background] Caglar B, Serin S, Yilmaz G, Torun A, Parlak I. The Impact of Treatment with Continuous Positive Airway Pressure on Acute Carbon Monoxide Poisoning. Prehosp Disaster Med. 2019 Dec;34(6):588-591. doi: 10.1017/S1049023X19005028. Epub 2019 Oct 22. PMID 31637993